CLINICAL TRIAL: NCT02038595
Title: The Norepinephrine Transporter: A Novel Target for Imaging Brown Adipose Tissue
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1008007284
Record Dates: First submitted 2014-01-10; First posted 2014-01-16 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2015-07

CONDITIONS: Brown Adipose Tissue
Keywords: brown adipose tissue
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy subjects (Experimental): Healthy subjects (male, female)
  Interventions: Radiation: PET imaging

INTERVENTIONS:
Radiation: PET imaging

SUMMARY:
This study seeks to assess a novel imaging technique to image brown adipose tissue utilizing the norepinephrine transporter.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30 yrs
* BMI < 24 kg/m2
* Caucasian

Exclusion Criteria:

* Current neuro-psychiatric illness
* substance abuse
* medical or neurological illnesses likely to affect physiology or anatomy, i.e., uncontrolled hypertension, cardiovascular disorders
* current pregnancy
* current breast feeding
* suicidal ideation or behavior
* use of medications which potentially affect NET binding within 2 weeks of the PET scans.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
detection of brown adipose tissue based on PET imaging | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Hwang JJ, Yeckel CW, Gallezot JD, Aguiar RB, Ersahin D, Gao H, Kapinos M, Nabulsi N, Huang Y, Cheng D, Carson RE, Sherwin R, Ding YS. Imaging human brown adipose tissue under room temperature conditions with (11)C-MRB, a selective norepinephrine transporter PET ligand. Metabolism. 2015 Jun;64(6):747-55. doi: 10.1016/j.metabol.2015.03.001. Epub 2015 Mar 5. PMID 25798999